CLINICAL TRIAL: NCT03172351
Title: Prospective Randomized Clinical Trial Comparing Extended Depth of Focus Intraocular Lenses With a Monofocal Intraocular Lens
Brief Title: EDoF IOLs vs Monofocal IOL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carl Zeiss Meditec AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AT LARA 829MP BER-401-16
Record Dates: First submitted 2017-05-24; First posted 2017-06-01 (Actual); Last update posted 2020-07-16 (Actual); Status verified 2020-07

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- EDoF1 (Experimental)
  Interventions: Device: Monofocal; Device: EDoF2
- Monofocal (Active Comparator)
  Interventions: Device: EDoF1; Device: EDoF2
- EDoF2 (Active Comparator)
  Interventions: Device: EDoF1; Device: Monofocal

INTERVENTIONS:
Device: EDoF1 — extended depth of focus IOL - EDoF1
  Arms: EDoF2; Monofocal
Device: Monofocal — Monofocal IOL
  Arms: EDoF1; EDoF2
Device: EDoF2 — Comparison EDoF2 IOL
  Arms: EDoF1; Monofocal

SUMMARY:
prospective, comparative (3 arms), randomized, multicentric clinical trial

ELIGIBILITY:
Inclusion Criteria:

* Patient informed of the consequences and constraints of the Clinical Investigational Plan and who has given his/her written informed consent;
* Patients of any gender, aged 50 to 80 years;
* Assured follow-up examinations;
* clinically significant bilateral cataract;

Exclusion Criteria:

* Patients unable to meet the limitations of the Clinical Investigational Plan or likely of non-cooperation during the trial;
* Patients whose freedom is impaired by administrative or legal order;
* Current participation in another drug or device investigation;
* Ocular disorders, other than cataract, that could potentially cause future acuity loss to a level of 0.20 logMAR (corrected) or worse in either eye
* Any anterior segment pathology that could significantly affect outcomes (e.g. chronic uveitis, iritis, corneal dystrophy, etc.)
* Pseudoexfoliations syndrome
* Pathologic miosis or Pharmacotherapy with miotic agent
* Keratoconus
* Chronic or recurrent uveitis
* Diabetic retinopathy
* Uncontrolled glaucoma and or IOP>24mmHg
* Choroidal hemorrhage,
* All kind of infections (acute ocular disease, external/internal infection, systemic infection)
* Traumatic cataract
* Aniridia
* Microphthalmia
* Amblyopia
* Degenerative visual disorders (e.g. macular degeneration, optic nerve atrophy, or retinal disorders)
* Patient expected to require retinal laser treatment before the end of the 4-6 months follow-up
* Previous intraocular and corneal surgery
* Expected postop. astigmatism greater than 1 D
* Any type of corneal disorder
* Systemic or ocular pharmacotherapy, which can impact the visual acuity,
* Former, current or foreseeable application of Tamsulosin or Silodosin (e.g. Flomax, Flomaxtra, Rapflo) ) which potentially can cause the floppy iris syndrome, insufficient dilation, or missing of appropriate iris structures which can compromise the standard procedure according to the investigator's opinion
* Patients who are unable to fixate for longer time (e.g. strabismus, nystagmus)
* Dementia
* pregnancy or lactation period for female patients

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2017-05-24 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Defocus curve measurement | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Zeiss Study Site, Freiburg im Breisgau, Germany

REFERENCES:
- [Derived] Reinhard T, Maier P, Bohringer D, Bertelmann E, Brockmann T, Kiraly L, Salom D, Piovella M, Colonval S, Mendicute J. Comparison of two extended depth of focus intraocular lenses with a monofocal lens: a multi-centre randomised trial. Graefes Arch Clin Exp Ophthalmol. 2021 Feb;259(2):431-442. doi: 10.1007/s00417-020-04868-5. Epub 2020 Sep 11. PMID 32915276